CLINICAL TRIAL: NCT03034070
Title: Whole-Body 3D T1-weighted MR Imaging Anatomical Sequences: GE mDixon vs FSE (View) Approaches in Prostate Cancer. Comparison of Diagnostic Performance of GE mDixon and FSE, for Bone and Node Staging in Patients With Prostate Cancer.
Brief Title: Whole-Body 3D T1-weighted MR Imaging Anatomical Sequences: GE mDixon vs FSE (View) Approaches in Prostate Cancer.
Acronym: TFE-TVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TFE TVE
Record Dates: First submitted 2017-01-17; First posted 2017-01-27 (Estimated); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Prostate Adenocarcinoma; Metastasis
Keywords: MRI; MRI sequences; prostate cancer; cancer; staging; bone metastasis; node metastasis
MeSH Terms: conditions — Neoplasm Metastasis; Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic performance 3D T1 (Other): A 3D T1-weighted GE mDixon MR imaging sequence will be added to the routine 3D T1-weighted FSE sequence. mDixon sub-sequences (Fat and In Phase) are compared to 3D T1-weighted FSE in terms of diagnostic accuracy for M and N staging in prostate cancer patients: Fat, In Phase, Fat+In Phase and the routine 3D T1 will be analyzed separately, blindly and randomly.
  Interventions: Diagnostic Test: Diagnostic performance 3D T1

INTERVENTIONS:
Diagnostic Test: Diagnostic performance 3D T1 — Although non-invasive, the prospective addition of a new MRI sequence to a routine MRI protocol is considered by our ethical committee as an "interventional" study.

SUMMARY:
This study will assess and compare the diagnostic performances and image quality of two WB 3D T1-weighted MR imaging sequences for bone and node staging in patients with prostate cancer : the FSE sequence and a gradient echo (GE) sequence. The latter sequence's main feature is its acquisition time of approximately 1.5 minutes, compared to 18 min for the FSE sequence, reducing the exam's acquisition time, patient discomfort and increasing machine availability.

DETAILED DESCRIPTION:
Whole-body (WB) magnetic resonance (MR) imaging has increasingly been used for the screening of bone and soft-tissue metastases in patients with prostate cancer (1). A limitation for its implementation is the 45-60 minutes duration of current WB MRI examinations. Conventional WB MR imaging studies consisted of anatomical two-dimensional (2D) T1-weighted and fat-suppressed fluid-sensitive (proton-density fat-saturated (PDFS) or short-tau inversion-recovery (STIR)) and of a functional diffusion-weighted imaging sequence. Recent research has confirmed the feasibility of replacing the 2D anatomical sequences by a single three-dimensional (3D) T1-weighted fast spin echo (FSE) sequence (2).

This study will assess and compare the diagnostic performances and image quality of two WB 3D T1-weighted MR imaging sequences for bone and node staging in patients with prostate cancer : the FSE sequence and a gradient echo (GE) sequence. The latter sequence's main feature is its acquisition time of approximately 1.5 minutes, compared to 18 min for the FSE sequence, reducing the exam's acquisition time, patient discomfort and increasing machine availability.

The aim of this study is to evaluate the feasibility of the replacement of the WB 3D T1-weighted FSE MR imaging sequence by the WB 3D T1-weighted GE MR imaging sequence.

ELIGIBILITY:
Inclusion Criteria:

* prostate cancer with high risk for metastases

Exclusion Criteria:

* contraindications to MRI

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-12; Primary Completion 2017-12-18 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic performances of 3D GE T1 sub-sequences | 3 months
  Sensitivity, sensibility, positive and negative Predictive Values (PV) will be calculated with the results of each reading, and compared.
  The physical parameters of the different techniques will also be compared (Signal-to-noise ratio, contrast-to-noise ratio, ...).

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lecouvet FE, El Mouedden J, Collette L, Coche E, Danse E, Jamar F, Machiels JP, Vande Berg B, Omoumi P, Tombal B. Can whole-body magnetic resonance imaging with diffusion-weighted imaging replace Tc 99m bone scanning and computed tomography for single-step detection of metastases in patients with high-risk prostate cancer? Eur Urol. 2012 Jul;62(1):68-75. doi: 10.1016/j.eururo.2012.02.020. Epub 2012 Feb 17. PMID 22366187
- [Result] Pasoglou V, Michoux N, Peeters F, Larbi A, Tombal B, Selleslagh T, Omoumi P, Vande Berg BC, Lecouvet FE. Whole-body 3D T1-weighted MR imaging in patients with prostate cancer: feasibility and evaluation in screening for metastatic disease. Radiology. 2015 Apr;275(1):155-66. doi: 10.1148/radiol.14141242. Epub 2014 Dec 15. PMID 25513855